CLINICAL TRIAL: NCT00921986
Title: Cleveland Clinic Arrhythmia Biospecimen Repository (Cleveland Clinic Arrhythmia BioBank)
Brief Title: Biospecimen Repository for Cardiac Arrhythmias at the Cleveland Clinic
Status: Recruiting | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Mina Chung, MD, Principal Investigator, The Cleveland Clinic
Other Study IDs: 09-176
Record Dates: First submitted 2009-06-15; First posted 2009-06-17 (Estimated); Last update posted 2025-09-10 (Actual); Status verified 2025-08

CONDITIONS: Arrhythmias, Cardiac
Keywords: genetics; biorepository; cardiac death; atrial fibrillation; ventricular fibrillation; ventricular tachycardia; supraventricular tachycardias; premature ventricular complexes; premature atrial complexes; atrioventricular and intraventricular blocks; sinus node dysfunction; syncope; vasovagal reactivity; postural orthostatic tachycardia syndrome
MeSH Terms: conditions — Arrhythmias, Cardiac; Death; Atrial Fibrillation; Ventricular Fibrillation; Tachycardia, Ventricular; Tachycardia, Supraventricular; Ventricular Premature Complexes; Atrial Premature Complexes; Sick Sinus Syndrome; Syncope; Postural Orthostatic Tachycardia Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biospecimens to be collected: DNA, RNA, plasma, & serum. Also tissue may be collected.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Arrhythmias: Patients with arrhythmias
- Control Subjects: Subjects that do not have a history of cardiac arrhythmias.

SUMMARY:
Biorepository of blood and or tissue samples from patients presenting with cardiac arrhythmia syndromes.

DETAILED DESCRIPTION:
The long-term objective of this research is to find genes and biologic pathways causing arrhythmia syndromes and other diseases or conditions. In order to achieve this objective the investigators will collect comprehensive phenotypic data and corresponding blood and/or tissue samples into a biorepository registry of patients, presenting for cardiac arrhythmia evaluation and/or treatment, and control subjects without arrhythmias. This biorepository will be composed of two parts: 1) An Arrhythmia Biorepository of blood and tissue from patients undergoing arrhythmia procedures, cardiac surgery, or inpatient or outpatient evaluations for arrhythmias, and 2) A Collaborative Sample Biorepository for de-identified samples and data from outside institutions and clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Male or female at least 18 years old
* Subjects with a history of or current cardiac arrhythmia, family members of subjects with cardiac arrhythmias, or no cardiac arrhythmia if a Control Subject.

Exclusion Criteria:

* Subjects previously enrolled in the Arrhythmia BioBank

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing arrhythmia procedures, cardiac surgery or inpatient or outpatient evaluations for arrhythmias at the Cleveland Clinic or from outside collaborative institutions or from other clinical trials.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2009-03 (Actual); Primary Completion 2035-12 (Estimated); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
Genetic variants associated with arrhythmias | Baseline
  Genome-wide association study of arrhythmias

CONTACTS AND LOCATIONS:
Overall Officials: Mina K. Chung, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No